CLINICAL TRIAL: NCT04707937
Title: Evaluation of a Brachytherapy Discharge Education Program (BrachDEP) to Improve Patient Care: A Randomized Control Trial
Brief Title: Evaluation of a Brachytherapy Discharge Education Program to Improve Patient Care
Acronym: BrachDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-5955
Record Dates: First submitted 2020-09-30; First posted 2021-01-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancer
Keywords: Brachytherapy; Vaginal Stenosis; Vaginal Toxicity; Online Education; Health Literacy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online education (Experimental): Participants will gain access to the online education modules in addition to receiving current standard of care education (pamphlets and one on one teaching with health care provider)
  Interventions: Other: Online education
- Regular standard of care education (Active Comparator): Participants only receive current standard of care education (pamphlets and one on one teaching with health care provider)
  Interventions: Other: Regular standard of care education

INTERVENTIONS:
Other: Online education — Access to online modules about brachytherapy education in addition to receiving regular standard of care education
  Arms: Online education
Other: Regular standard of care education — Access only to regular standard of care education
  Arms: Regular standard of care education

SUMMARY:
Although brachytherapy is an effective treatment modality for gynecological cancer, a significant proportion of patients develop late treatment-related vaginal toxicity, negatively impacting their quality of life and limiting recurrent disease detection by preventing adequate clinical examination during the post-treatment surveillance period. Consistent with the literature, results from a study at Princess Margaret revealed that current vaginal toxicity management education and training may be inadequate. The investigators seek to implement and evaluate a new online brachytherapy discharge education program (BrachDEP) to support patient engagement in self-management.

DETAILED DESCRIPTION:
Background:

Brachytherapy is a type of radiation therapy used to treat patients with gynecological cancers. Brachytherapy delivers radiation to cancerous tissue by inserting or placing the radiation next to the target tissue. A common side effect that develops as a result of repeated brachytherapy is fibrosis, a thickening and hardening of tissue, as well as narrowing of the vagina, known as vaginal stenosis. To reduce the impact of vaginal stenosis, vaginal dilation is recommended upon discharge of brachytherapy. Vaginal dilation involves the insertion of a smooth plastic tube into the vagina 3 to 4 times per week. Despite the benefits of vaginal dilation, use of vaginal dilators is low among patients following brachytherapy. This poor adherence to vaginal dilator use may be due to embarrassment, discomfort, and lack of awareness of the benefits to patients.

Objective:

The primary objective of this study is to evaluate the whether an online brachytherapy discharge education program increases patient satisfaction with education and care. Secondary objectives are to determine whether the online education program increases patient quality of life, improves vaginal dilator compliance and reduces rates of vaginal stenosis post-treatment.

Methods:

The research team will use a randomized, controlled trial study design. The impact of the online education program will be identified by comparing the outcomes of participants in the intervention arm against those patients in the control arm. Participants will be recruited and randomized to one of two arms that will determine whether they will receive the education intervention.

Significance The results from this study will be used to improve the brachytherapy discharge education program.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive brachytherapy for treatment of gynecologic cancer at Princess Margaret Cancer Centre.
* Able to provide written informed consent
* Able to read and write in English
* > 18 years of age

Exclusion Criteria:

* Not receiving brachytherapy treatment

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecological cancer patients receiving brachytherapy treatment
Enrollment: 150 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction with access to education (CBI) | 1 year
  To determine whether the online brachytherapy discharge education program increases patient satisfaction with education and care.
  CBI: Cancer Behavioural Inventory Brief min score: 12 max score: 108 higher scores indicates greater coping efficacy
Patient Satisfaction with access to education (EQ-5D-5L) | 1 year
  To determine whether the online brachytherapy discharge education program increases patient satisfaction with education and care.
  Health Status min value set: 11111 max value set: 55555 lower value set indicates better health
  min score: 0% max score: 100% higher percentage indicates best possible health
Patient Satisfaction with access to education (EORTC-QOL) | 1 year
  To determine whether the online brachytherapy discharge education program increases patient satisfaction with education and care.
  Quality of Life min score: 1 max score 100 higher score indicates higher level of functioning
Patient Satisfaction with access to education (SVQ) | 1 year
  To determine whether the online brachytherapy discharge education program increases patient satisfaction with education and care.
  The sexual function vaginal changes questionnaire higher scores indicate better overall sexual functioning
Patient Satisfaction with access to education (PS-CaTE) | 1 year
  To determine whether the online brachytherapy discharge education program increases patient satisfaction with education and care.
  Patient Satisfaction with Cancer Treatment Education min score = 1 max score = 5 higher score indicates greater satisfaction with information

SECONDARY OUTCOMES:
Rates of vaginal stenosis | 1 year
  To determine whether the online brachytherapy discharge education program:
  1. Increases patient quality of life
  2. Improves vaginal dilator compliance
  3. Reduces rates of vaginal stenosis for gynecological cancer patients post treatment
  Will be measured by tracking dilator compliance diary and measuring vaginal toxicity at baseline and 1-year post treatment (Vaginal Morbidity at Gynecological Examination)
  Higher scores indicate lower vaginal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Janet Papadakos, PhD, MEd, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No